CLINICAL TRIAL: NCT04323800
Title: Convalescent Plasma to Stem Coronavirus: A Randomized, Blinded Phase 2 Study Comparing the Efficacy and Safety Human Coronavirus Immune Plasma (HCIP) vs. Control (SARS-CoV-2 Non-immune Plasma) Among Adults Exposed to COVID-19
Brief Title: Convalescent Plasma to Stem Coronavirus (CSSC-001)
Acronym: CSSC-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00245634
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Results first posted 2022-04-22 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Coronavirus; Convalescence
Keywords: COVID-19
MeSH Terms: conditions — Coronavirus Infections; Convalescence; COVID-19

STUDY DESIGN:
Intervention Model Description: 1:1 ratio
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- High titer anti-SARS-CoV-2 plasma (Experimental): Participants with High titer anti-SARS-CoV-2 plasma.
  Interventions: Biological: Anti- SARS-CoV-2 Plasma
- SARS-CoV-2 non-immune plasma (Active Comparator): Participants with SARS-CoV-2 non-immune plasma.
  Interventions: Biological: SARS-CoV-2 non-immune Plasma

INTERVENTIONS:
Biological: Anti- SARS-CoV-2 Plasma — SARS-CoV-2 convalescent plasma (1 unit; ~200-250 mL collected by pheresis from a volunteer who recovered from COVID-19 disease and has SARS-CoV-2 antibody titers ≥ 1:320
  Arms: High titer anti-SARS-CoV-2 plasma
Biological: SARS-CoV-2 non-immune Plasma — Normal human plasma collected prior to December 2019
  Arms: SARS-CoV-2 non-immune plasma

SUMMARY:
Evaluate the efficacy of treatment with high-titer Anti- SARS-CoV-2 plasma versus control (SARS-CoV-2 non-immune plasma) in subjects exposed to Coronavirus disease (COVID-19) at day 28.

DETAILED DESCRIPTION:
This randomized, controlled, double-blinded phase 2 trial will assess the efficacy and safety of Anti- SARS-CoV-2 convalescent plasma as prophylaxis following exposure to COVID-19 (as defined in the inclusion criteria). Adults 18 years of age and older with high risk exposure as defined by CDC may participate. A total of 500 eligible subjects will be randomized in a 1:1 ratio to receive either high titer anti-SARS-CoV-2 plasma or control (SARS-CoV-2 non-immune plasma).

ELIGIBILITY:
Inclusion Criteria

1. Subjects must be 18 years of age or older
2. Close contact exposure (as defined by CDC guidelines) to person with COVID-19 within 96 hours of randomization (and 120 hours of receipt of plasma)

Exclusion Criteria

1. Receipt of any blood product in past 120 days.
2. Medical, psychiatric,cognitive illness or recreational drug/alcohol use that in the opinion of the principal investigator, would affect subject safety and/or compliance.
3. Symptoms consistent with COVID-19 infection (fevers, acute onset cough, shortness of breath) at time of screening.
4. Laboratory evidence of COVID-19 infection at time of screening.
5. History or known laboratory evidence of previous COVID-19 infection.
6. History of prior reactions to transfusion blood products.
7. Inability to complete therapy with the study product within 24 hours after randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2021-04-22 (Actual); Study Completion 2021-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shmuel Shoham, MD, Principal Investigator — Johns Hopkins University
Locations (25):
- United States (25):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Center for American Indian Health - Whiteriver Office, Whiteriver, Arizona
  - University of California, San Diego, La Jolla, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Irvine Health, Orange, California
  - Western Connecticut Health Network, Danbury Hospital, Danbury, Connecticut
  - Western Connecticut Health Netowrk, Norwalk Hospital, Norwalk, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Miami, Coral Gables, Florida
  - University of Miami Clinical Translational Research Site, Miami, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
  - Anne Arundel Medical Center, Annapolis, Maryland
  - The Johns Hopkins University, Baltimore, Maryland
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Center for American Indian Health - Gallup Office, Gallup, New Mexico
  - Center for American Indian Health - Shiprock Office, Shiprock, New Mexico
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Lifespan/BrownUniversity (Rhode Island Hospital), Providence, Rhode Island
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - The University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Sharing is governed by Johns Hopkins University Institutional Guidelines

REFERENCES:
- [Derived] Shoham S, Bloch EM, Casadevall A, Hanley D, Lau B, Gebo K, Cachay E, Kassaye SG, Paxton JH, Gerber J, Levine AC, Naeim A, Currier J, Patel B, Allen ES, Anjan S, Appel L, Baksh S, Blair PW, Bowen A, Broderick P, Caputo CA, Cluzet V, Cordisco ME, Cruser D, Ehrhardt S, Forthal D, Fukuta Y, Gawad AL, Gniadek T, Hammel J, Huaman MA, Jabs DA, Jedlicka A, Karlen N, Klein S, Laeyendecker O, Lane K, McBee N, Meisenberg B, Merlo C, Mosnaim G, Park HS, Pekosz A, Petrini J, Rausch W, Shade DM, Shapiro JR, Singleton JR, Sutcliffe C, Thomas DL, Yarava A, Zand M, Zenilman JM, Tobian AAR, Sullivan DJ. Transfusing Convalescent Plasma as Post-Exposure Prophylaxis Against Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection: A Double-Blinded, Phase 2 Randomized, Controlled Trial. Clin Infect Dis. 2023 Feb 8;76(3):e477-e486. doi: 10.1093/cid/ciac372. PMID 35579509
- [Derived] Shoham S, Bloch EM, Casadevall A, Hanley D, Lau B, Gebo K, Cachay E, Kassaye SG, Paxton JH, Gerber J, Levine AC, Currier J, Patel B, Allen ES, Anjan S, Appel L, Baksh S, Blair PW, Bowen A, Broderick P, Caputo CA, Cluzet V, Cordisco ME, Cruser D, Ehrhardt S, Forthal D, Fukuta Y, Gawad AL, Gniadek T, Hammel J, Huaman MA, Jabs DA, Jedlicka A, Karlen N, Klein S, Laeyendecker O, Lane K, McBee N, Meisenberg B, Merlo C, Mosnaim G, Park HS, Pekosz A, Petrini J, Rausch W, Shade DM, Shapiro JR, Singleton JR, Sutcliffe C, Thomas DL, Yarava A, Zand M, Zenilman JM, Tobian AAR, Sullivan D. Randomized controlled trial transfusing convalescent plasma as post-exposure prophylaxis against SARS-CoV-2 infection. medRxiv [Preprint]. 2021 Dec 14:2021.12.13.21267611. doi: 10.1101/2021.12.13.21267611. PMID 34931202

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Titer Anti-SARS-CoV-2 Plasma | SARS-CoV-2 Non-immune Plasma
Started | 87 | 93
Completed | 81 | 87
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Incomplete transfusion | 1 | 0
Not completed — Other | 0 | 1
Not completed — Positive RT-PCR at transfusion | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Titer Anti-SARS-CoV-2 Plasma | SARS-CoV-2 Non-immune Plasma | Total
Number analyzed (Participants) | 87 | 93 | 180
Age, Continuous [Median (Full Range); unit: years] | 48 [19 to 82] | 46 [18 to 91] | 48 [18 to 91]
Age, Customized [Count of Participants; unit: Participants]
  18 - 34 years | 18 | 26 | 44
  35 - 44 years | 19 | 18 | 37
  45 - 54 years | 22 | 19 | 41
  55 - 64 years | 14 | 16 | 30
  >/=65 years | 14 | 14 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 81
  Male | 46 | 53 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 16 | 31
  Not Hispanic or Latino | 72 | 77 | 149
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 7 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 6 | 10
  White | 80 | 78 | 158
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
BMI [Count of Participants; unit: Participants] — Body Mass Index (BMI) of participants (Kg/m^2).
  Participants
    <18 | 2 | 0 | 2
    18-24.9 | 23 | 34 | 57
    25-29.9 | 30 | 14 | 44
    30-34.9 | 10 | 16 | 26
    35-39.9 | 6 | 11 | 17
    >/=40 | 3 | 5 | 8
    Missing | 13 | 13 | 26
Number of people in household [Count of Participants; unit: Participants]
  1 | 18 | 26 | 44
  2 | 19 | 21 | 40
  3 | 17 | 15 | 32
  4 | 17 | 10 | 27
  >/=5 | 12 | 17 | 29
  Missing | 4 | 4 | 8
Number of household COVID-19 positives [Count of Participants; unit: Participants]
  1 | 54 | 54 | 108
  2 | 8 | 5 | 13
  3 | 1 | 3 | 4
  >/=4 | 0 | 1 | 1
  Missing | 24 | 30 | 54
Median time from last exposure to transfusion [Median (Inter-Quartile Range); unit: hours] | 2 [1 to 4] | 3 [1 to 4] | 3 [1 to 4]
Days from last exposure to transfusion [Count of Participants; unit: Participants]
  0 | 7 | 7 | 14
  1 | 24 | 16 | 40
  2 | 12 | 14 | 26
  3 | 11 | 17 | 28
  4 | 12 | 16 | 28
  >/=5 | 7 | 9 | 16
  Missing | 9 | 9 | 18
  Not transfused | 5 | 5 | 10
Cancer Status [Count of Participants; unit: Participants]
  Active cancer | 1 | 1 | 2
  Active cancer on chemotherapy | 0 | 1 | 1
  Cancer in remission | 6 | 5 | 11
  Leukemia/Lymphoma | 2 | 6 | 8
  No cancer | 78 | 80 | 158
Cardiac condition [Count of Participants; unit: Participants]
  Arrhythmia | 2 | 1 | 3
  Atrial fibrillation, on anticoagulant | 1 | 0 | 1
  Cardiomyopathy | 1 | 0 | 1
  Coronary artery disease | 1 | 3 | 4
  Myocardial infarction | 0 | 2 | 2
  No cardiac condition | 82 | 87 | 169
Immunologic condition [Count of Participants; unit: Participants]
  Allergic rhinitis | 12 | 10 | 22
  Inflammatory bowel disease | 0 | 3 | 3
  HIV, on antiretroviral treatment | 4 | 6 | 10
  Psoriasis | 2 | 0 | 2
  Immunosuppression or on other immune modulator | 1 | 0 | 1
  No immunologic condition | 68 | 74 | 142
Metabolic condition [Count of Participants; unit: Participants]
  Diabetes Mellitus | 6 | 5 | 11
  Vitamin D deficiency | 1 | 1 | 2
  No metabolic condition | 80 | 87 | 167
Respiratory condition [Count of Participants; unit: Participants]
  Asthma | 4 | 5 | 9
  Chronic Bronchitis | 0 | 2 | 2
  Chronic sinusitis | 0 | 1 | 1
  Cough | 1 | 1 | 2
  Pulmonary fibrosis | 0 | 1 | 1
  Pulmonary hypertension | 1 | 1 | 2
  No respiratory condition | 81 | 82 | 163
Tobacco use status [Count of Participants; unit: Participants]
  Current tobacco user | 2 | 1 | 3
  Past tobacco user | 1 | 4 | 5
  No tobacco use | 84 | 88 | 172

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Treatment at Day 28 as Assessed by Number of Participants Who Develop SARS-Cov-2 Infection
Description: Comparison of proportions of cumulative incidence of development of SARS-Cov-2 infection (symptoms compatible with infection and/or + molecular testing) regardless of disease severity, following high-titer Anti- SARS-CoV-2 plasma versus control (SARS-CoV-2 non-immune plasma) in subjects exposed to COVID-19.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | High Titer Anti-SARS-CoV-2 Plasma | SARS-CoV-2 Non-immune Plasma
Number analyzed (Participants) | 81 | 87
Participants | 12 | 13
Statistical Analysis 1: Comparison: High Titer Anti-SARS-CoV-2 Plasma vs SARS-CoV-2 Non-immune Plasma; Test type: Superiority; p = 0.42, Restricted Mean Survival Test statistic — One-sided p-value; Risk Difference (RD) = 0.01

2. Primary Outcome: Safety of Treatment With High-titer Anti- SARS-CoV-2 Plasma Versus Control as Assessed by Number of Participants With "Serious Adverse Events"
Description: Number of participants with serious adverse events categorized as either severe infusion reactions or Acute Respiratory Distress Syndrome during the study period.
Time Frame: Up to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | High Titer Anti-SARS-CoV-2 Plasma | SARS-CoV-2 Non-immune Plasma
Number analyzed (Participants) | 81 | 87
Participants | 0 | 1
Statistical Analysis 1: Comparison: High Titer Anti-SARS-CoV-2 Plasma vs SARS-CoV-2 Non-immune Plasma; Test type: Superiority; p = 0.67, Chi-squared; Risk Difference (RD) = -5, 95% CI 2-sided [-31 to 19]

3. Primary Outcome: Safety of Treatment With High-titer Anti- SARS-CoV-2 Plasma Versus Control as Assessed by Cumulative Incidence of Grade 3 and 4 Adverse Events
Description: Cumulative incidence of grade 3 and 4 adverse events during the study period evaluated as events per 100 person-years will be used to assess safety of the intervention.
Time Frame: Up to Day 28
Measure: Number (95% Confidence Interval); unit: Events per 100 person-years
Arm/Group | High Titer Anti-SARS-CoV-2 Plasma | SARS-CoV-2 Non-immune Plasma
Number analyzed (Participants) | 81 | 87
Events per 100 person-years | 23 [6 to 61] | 70 [37 to 120]
Statistical Analysis 1: Comparison: High Titer Anti-SARS-CoV-2 Plasma vs SARS-CoV-2 Non-immune Plasma; Test type: Superiority; p = 0.06, Chi-squared; Risk Difference (RD) = -47, 95% CI 2-sided [-100 to 2]

4. Secondary Outcome: Number of Participants With Severe Disease
Description: Number of participants with severe disease between the anti-SARS-CoV-2 convalescent plasma and control groups. Severity of disease will be measured using the number of participants with any of the disease severity categories below:
  1. Death
  2. Requiring mechanical ventilation and/or in ICU
  3. non-ICU hospitalization, requiring supplemental oxygen
  4. non-ICU hospitalization, not requiring supplemental oxygen
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | High Titer Anti-SARS-CoV-2 Plasma | SARS-CoV-2 Non-immune Plasma
Number analyzed (Participants) | 81 | 87
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Within 28 days
Description: Adverse events were evaluated among those transfused and not SARS Cov-2 positive at baseline. Adverse Events were monitored/assessed without regard to the specific Adverse Event Term.
Arm/Group | High Titer Anti-SARS-CoV-2 Plasma | SARS-CoV-2 Non-immune Plasma
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/87
Serious Adverse Events (participants affected / at risk) | 4/81 | 14/87
Other Adverse Events (participants affected / at risk) | 24/81 | 44/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Titer Anti-SARS-CoV-2 Plasma (N=81) | SARS-CoV-2 Non-immune Plasma (N=87)
Severe transfusion reaction (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Grade 3 or 4 adverse events (General disorders) | 4 (4) | 13 (13)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Titer Anti-SARS-CoV-2 Plasma (N=81) | SARS-CoV-2 Non-immune Plasma (N=87)
Non-serious adverse events (General disorders) | 24 (24) | 44 (44)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/00/NCT04323800/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT04323800/SAP_001.pdf
  • Informed Consent Form (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT04323800/ICF_002.pdf